CLINICAL TRIAL: NCT06309017
Title: Pre-operative Nutrition for Elective Resection Surgery in Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-01243
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition specialist (Experimental): Participants will be assigned to this arm if the subject is determined malnourished. They will be sent to a nutrition specialist for a nutrition focused visit and will be provided standard of care intervention prior surgery.
  Interventions: Other: Nutrition specialist; Dietary Supplement: Ensure Surgery Immunonutrition shakes
- Standard of Care (Active Comparator): Participants that show no signs of malnutrition will be assigned to this arm. The subject will be provided with education and schedule of Ensure® Surgery Immunonutrition shakes for prior to surgery as per standard of care.
  Interventions: Dietary Supplement: Ensure Surgery Immunonutrition shakes

INTERVENTIONS:
Other: Nutrition specialist — Nutrition specialist to help improve nutritional status by diet, oral nutrition supplements or parenteral nutrition.
  Arms: Nutrition specialist
Dietary Supplement: Ensure Surgery Immunonutrition shakes — All study subjects, including subjects without malnutrition, will be given the Ensure Surgery Immunonutrition Shakes for prior to surgery as per standard of care. All subjects will also receive additional shakes starting as an inpatient when diet is advanced.

SUMMARY:
This study aims to determine if improved risk stratification tools and interventions to mitigate malnutrition reduce postoperative risk in patients undergoing elective or emergent resection surgery for inflammatory bowel disease (IBD), and if adding immune modulation nutrition improves surgical outcomes. The primary objective is to assess whether preoperative malnutrition screening and intervention minimize postoperative complications. The secondary objective is to evaluate whether immune modulation nutrition in the peri-operative period decreases length of stay and major complications.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent
2. Aged 18 years of age or older
3. Confirmed diagnosis of inflammatory bowel disease
4. Scheduled for disease-related intestinal resection at NYU Langone Health

Exclusion Criteria:

1. No current diagnosis of inflammatory bowel disease
2. Age less than 18
3. Not proficient (able to read and answer questions) in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 30 days post-surgery
  From the time the patient is admitted at hospital for surgery until the patient is discharged.
Proportion of patients who experienced postoperative major complications | Visit 3 (30 days post-surgery)
  Major complications include infection, bleeding (requiring blood transfusion or requiring intervention), cardiac event (myocardial infarction, arrhythmia, and cardiac arrest), stroke, acute kidney injury (increase in serum creatinine of ≥0.3 mg/dL from baseline or ≥1.5 times baseline), venous thromboembolism, reoperation, readmission, and need for ICU-level care. The outcome measure will be obtained from the electronic health record (EHR).

SECONDARY OUTCOMES:
Proportion of patients who participated in a nutritional intervention program before surgery | Visit 3 (30 days post-surgery)
Proportion of patients who participated in a nutritional intervention program after surgery | Visit 3 (30 days post-surgery)
Number of nutritional shakes completed | Visit 3 (30 days post-surgery)
Percentage of nutritional shakes completed overall | Visit 3 (30 days post-surgery)
Percentage of nutritional shakes completed pre-surgery | One day prior to surgery
  Subject will be called the day prior to surgery to determine the number of shakes consumed by patient.
Percentage of nutritional shakes completed post-surgery | One week post surgery
  One week after surgery, a phone call will follow to determine how many shakes subject consumed.
Proportion of patients who experienced any postoperative complications | Visit 3 (30 days post-surgery)
Proportion of patients with 30 day readmission | Up to 30 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Katz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Jennifer.katz@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Jennifer.katz@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.